CLINICAL TRIAL: NCT05263726
Title: The Effect of a Disease Self-management Program Through a Mobile Applications for Patients With Hypertension
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taipei University of Nursing and Health Sciences (Other)
Collaborators: Cardinal Tien Hospital (Other)
Responsible Party: Principal Investigator, Mei-Chen Lee, RN, PhD, Associate Professor, National Taipei University of Nursing and Health Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: CTH-109-3-1-062
Record Dates: First submitted 2022-02-14; First posted 2022-03-03 (Actual); Last update posted 2023-03-23 (Actual); Status verified 2023-03

CONDITIONS: Hypertension; Self-management; Mobile Applications
Keywords: mobile applications; hypertension; disease self-management program; mental health; self-management; quality of life
MeSH Terms: conditions — Hypertension; Psychological Well-Being

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DSMP through a mobile applications (Experimental): This interventional divided the disease self-management program manual for patients with hypertension into 4 units, including: Unit 1: hypertension brief introduction and complications. Unit 2: dietary precautions for patients with hypertension. Unit 3: medication treatments for patients with hypertension. Unit 4: the content included stress management (emotional control, spiritual support) of patients with hypertension. The experimental group received the mobile apps educational program for at least 30 minutes each session and at least once every two days. After two weeks and six weeks, a follow-up telephone interview helped to strengthen the health self-management self-confidence. The researcher used the back office administration at the computer end to observe how the experimental group operated and used the mobile devices. The effect of interventions was then evaluated after three months when the patients returned.
  Interventions: Behavioral: DSMP through a Mobile Applications
- Usual Care (No Intervention): Routine care

INTERVENTIONS:
Behavioral: DSMP through a Mobile Applications — This interventional divided the disease self-management program manual for patients with hypertension into 4 units, including: Unit 1: hypertension brief introduction and complications. Unit 2: dietary precautions for patients with hypertension. Unit 3: medication treatments for patients with hypertension. Unit 4: the content included stress management (emotional control, spiritual support) of patients with hypertension. The experimental group received the mobile apps educational program for at least 30 minutes each session and at least once every two days. After two weeks and six weeks, a follow-up telephone interview helped to strengthen the health self-management self-confidence. The researcher used the back office administration at the computer end to observe how the experimental group operated and used the mobile devices. The effect of interventions was then evaluated after three months when the patients returned.
  Arms: DSMP through a mobile applications

SUMMARY:
Hypertension is a major cause of death worldwide. Patients should adjust their lifestyle and learn how to maintain a balance between self-management of a disease and their daily livelihood. Knowledge is networked, mobile devices can be used as a way of health education. The purpose of this study is to evaluation the effectiveness of the disease self-management program through a mobile applications for patients with hypertension. Statistical analyses was used analysis of covariance for checking the effect of interventions. Through the calculation by a statistical power analysis formula, the study takes 70 samples and divides them into a control group (usual care) and an experimental group (disease self-management program through a mobile applications) by the single blind randomized controlled trial, whereby each groups has 35 samples. The first step investigate the physiological indicators, mental health, self-management, quality of life of the patients. For the experimental group, after the pre-test the study set up a health guide for the disease self-management program with a mobile applications. The experimental group received the mobile apps educational program for at least 30 minutes each session and at least once every two days. After two weeks and six weeks, a follow-up telephone interview helped to strengthen the health self-management self-confidence. The effect of interventions was then evaluated after three months when the patients returned. Therefore, the self-management of a disease can be improved and patients will learn to live in harmony with hypertension by improving their mental health, self-management, and quality of life.

DETAILED DESCRIPTION:
Due to the aging population and the advancement of medical science and technology, people's lives have been extended longer in years, but at the same time the prevalence rate of chronic diseases is increasing. Hypertension may cause several complications, resulting in abnormal organs either chronically or deadly. Patients should adjust their lifestyle and learn how to maintain a balance between self-management of a disease and their daily livelihood. Knowledge is networked, mobile devices can be used as a way of health education. Therefore, this research builds a disease self-management program through a mobile applications that runs in accordance with expert validity, so as to effectively control hypertension and avoid its complications. SPSS/Windows 22.0 helped with filing and statistical analyses, and analysis of covariance (ANCOVA) was used for checking the effect of interventions. Through the calculation by a statistical power analysis formula, the study takes 70 samples and divides them into a control group (usual care) and an experimental group (disease self-management program through a mobile applications) by the single blind random control trial, whereby each groups has 35 subjects. The first step tests the physiological indicators, mental health, self-management, and quality of life of the patients. For the experimental group, after the pre-test the study set up a health guide for the disease self-management program with a mobile applications. The experimental group received the mobile apps educational program for at least 30 minutes each session and at least once every two days. After two weeks and six weeks, a follow-up telephone interview helped to strengthen the health self-management self-confidence. The effect of interventions was then evaluated after three months when the patients returned. The findings are expected to effectively control patients' hypertension in Taiwan after completing the research plan. Therefore, the self-management of a disease can be improved and patients will learn to live in harmony with hypertension by improving their mental health, self-management, and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Hypertension Disease
* A clear state of consciousness and without diagnosis of mental illness
* Can communicate in Chinese and Taiwanese and are willing to participate in this study
* Age 18 years old the above

Exclusion Criteria:

* Cognitive dysfunction who are unable to understand the questionnaire
* Mental illness (severe depression, schizophrenia) reported in the medical records.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2022-02-08 (Actual); Primary Completion 2023-01-30 (Actual); Study Completion 2023-01-30 (Actual)

PRIMARY OUTCOMES:
The Partner in Health Scale (PIH) | Change from Baseline Disease Self-management at 3 months.
  This scale is a generic tool that was developed for measuring self-management knowledge and behaviors in patients with chronic illnesses (Battersby et al., 2003). Original scale includes 11 items, contains five properties. The internal consistency reliability Cronbach's α value of this scale is .88. Then redefinition the six major principles of chronic condition self-management including disease knowledge, adherence to a treatment plan made in accordance with the healthcare provider, playing an active role in the decision-making process, awareness of warning symptoms and their management, coping with the effects the of the chronic illness in relation to the physical, mental and social aspects of life and practice of a healthy lifestyle. The PIH scale is a self-report questionnaire that includes 12 items, which are answered using 9-point Likert-type scales (from 0 "very poor" to 8 "very well"). The total score ranges from 0 to 96, 0 representing poor self-management and 96 representing

SECONDARY OUTCOMES:
World Health Organization-5 Well Being Index (WHO-5) | Change from Baseline Mental Health at 3 months.
  This scale is a 5-item questionnaire. The scoring included 0 point (at no time), representing the worst to 5 points (all of the time), representing the best. The total score ranges from 0 to 25 points. Patients whose total score is lower than 13 points or whose answer to any of the 5 items is 0 to 1 point are recommended to receive the test of severe depression scale or review a face-to-face interview with a psychologist to check whether they meet the medical diagnosis of depression. The internal consistency reliability Cronbach's α value of this scale is .87. The test-retest reliability of this scale in Germany and Japan is Cronbach's α .90 (Saipanish, Lotrakul, & Sumrithe, 2009). The internal consistency reliability Cronbach's α value of this scale in Taiwan is Cronbach's α .89 (Lee et al., 2021)
Medical Outcome Study Short Form-12 (MOS SF-12) | Change from Baseline quality of life at 3 months.
  Both the SF-12 and SF-36 quality of life scales are derived from the Medical Outcomes Study (MOS). SF-12 was finalized in 1994, with a total of 12 questions in two dimensions, PCS and MCS, which were four reverse questions (questions 1, 5, 6a, and 6b) that needed to be scored in reverse first. As the measuring scale and scoring method of each question are different, it must be converted to the order of 0-100 points, where 100 points indicates the best condition. The total score of all questions are divided by 12 to obtain the total score of the scale, which ranges from 0 to 120 points, the higher the score, the better the quality of life of the patients. In 2021, Chen et al. (2021) used the SF-12 scale to measure patients with hypertensive nephropathy. The results showed that the internal consistency Cronbach's α values of SF-12 were 0.88, 0.87, and 0.87, respectively, for the overall quality of life, quality of life in the PCS, and quality of life in the MCS.

CONTACTS AND LOCATIONS:
Overall Officials: Mei-Chen Lee, PhD, Principal Investigator — National Taipei University of Nursing and Health Sciences
Locations (1):
- Cardinal Tien Hospital, New Taipei City, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chen CW, Lu YY, Lin LJ, Liu JH, Lee MC, Wu SV. Using a Mobile Application Disease Self-management Program to Promote Blood Pressure Control and Quality of Life in Patients With Hypertension. Comput Inform Nurs. 2025 Mar 14. doi: 10.1097/CIN.0000000000001296. Online ahead of print. PMID 40084962
- See also: Mobile health applications for the management of primary hypertension: A multicenter, randomized, controlled trial. — https://doi.org/10.1097/MD.0000000000019715
- See also: The effectiveness of electronic health interventions on blood pressure control, self-care behavioral outcomes and psychosocial well-being in patients with hypertension: A systematic review and meta-analysis. — https://doi.org/10.1016/j.ijnurstu.2018.11.007